CLINICAL TRIAL: NCT01980862
Title: Blood Collection From Heart Failure Patients to Evaluate for Galectin-3 Measurement Differences Using Various Collection Tubes
Status: Completed | Type: Observational
Sponsor: Fujirebio Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FDI-83
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: To Measure Galectin-3 in Heart Failure Patients on Commercial Platforms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Heart Failure patients: No interventions for this study. Blood draw provided by patients.

SUMMARY:
Single-site blood collection investigation.

DETAILED DESCRIPTION:
45 Heart Failure patients will be recruited. Patients will provide a one-time blood sample specimen collection. Theses samples will be de-identified and provided for measurement of Galectin-3 on commercial platforms.

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure patients New York Heart Association class able to provide (4) collection tube types Subjects > 18 years old All subjects must provide informed consent and associated documentation

Exclusion Criteria:

* Subjects that cannot tolerate blood withdrawal of 4 specimens collection tube tubes (approximately 40 mLs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45 matched door serum and plasma. Samples set collected form individual Heart Failure patients for galecin-3 measurements
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Obtain 45 matched donor serum and plasma samples sets collected from Heart Failure patients for galectin-3 measurements | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Christenson, MD, Principal Investigator — Universtiy of Maryland School of Medicine
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States